CLINICAL TRIAL: NCT03127215
Title: A Randomized Phase-2 Study of Trabectedin/Olaparib Compared to Physician's Choice in Subjects With Previously Treated Advanced or Recurrent Solid Tumors Harboring DNA Repair Deficiencies
Brief Title: Study of Olaparib/Trabectedin vs. Doctor's Choice in Solid Tumors
Acronym: NCT-PMO-1603
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: AstraZeneca (Industry); PharmaMar (Industry); German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2017-0417
Record Dates: First submitted 2017-03-31; First posted 2017-04-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-08

CONDITIONS: Cancers With DNA Repair-Deficiency
MeSH Terms: interventions — olaparib; Trabectedin

STUDY DESIGN:
Intervention Model Description: randomized
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm E: Olaparib / Trabectedin (Experimental): Olaparib / Trabectedin
  Interventions: Drug: Olaparib; Drug: Trabectedin
- Arm C: Physician's choice (Other): Physician's choice
  Interventions: Drug: Physician's choice

INTERVENTIONS:
Drug: Olaparib — Olaparib 150 mg tablet
  Arms: Arm E: Olaparib / Trabectedin
Drug: Physician's choice — treatment according to current guidelines
  Arms: Arm C: Physician's choice
Drug: Trabectedin — Trabectedin 1.1mg/m² infusional solution
  Arms: Arm E: Olaparib / Trabectedin

SUMMARY:
Evaluation of the efficacy of the combination of olaparib and trabectedin in adult patients with locally advanced/metastatic solid tumors that failed standard treatment and whose molecular sequencing tumor profiles show homologous recombination repair (HRR) defects. The primary objective is to show superior disease control rate in patients with HRR-deficient tumors treated with olaparib and trabectedin compared to treatment according to current guidelines (physician's choice). This trial aims to establish whether the PARP-dependency of HRR-deficient tumors across entities can be exploited for therapeutic benefit.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Progressive locally advanced or metastatic malignancy
* Prior administration of standard treatment for primary and relapsed malignancy
* Eastern Cooperative Oncology Group Performance Status ≤1
* Patients with central venous access device in place (central venous catheter or porta-cath)
* Age ≥18 and ≤70 years
* Identification of defective DNA repair via HR
* Adequate bone marrow, renal, and hepatic function
* Hemoglobin ≥10 g/dl
* Neutrophil count ≥1,500/mm3
* Platelet count ≥100,000/µl
* Bilirubin ≤1.5 x upper limit of normal (ULN)
* ALT and AST ≤2.5 x ULN (≤5 x ULN in patients with hepatic tumor involvement)
* Alkaline phosphatase ≤2.5 x ULN
* PT-INR/PTT ≤1.5 x ULN
* Albumin ≥25 g/l
* Creatine kinase ≤2.5 x ULN
* Serum creatinine 1.5 mg/dl or creatinine clearance 51 ml/min

Main Exclusion Criteria:

* Hematological malignancies and primary brain tumors.
* Concurrent treatment in another interventional clinical trial
* Prior treatment with PARP Inhibitors
* Patients with platinum-refractory disease, defined as progressive disease during or immediately after treatment with platinum based chemotherapy
* Persistent toxicity (> Grade 2 according to CTCAE 5.0)
* Dementia or significant impairment of cognitive state
* History of HIV infection
* Clinical signs of active infection (>Grade 2 according to CTCAE 4.03)
* History of viral hepatitis (HBV or HCV)
* Epilepsy requiring pharmacologic treatment
* Pregnancy
* Major surgical intervention 4 weeks prior to study inclusion
* Known hypersensitivity to any of the study drugs
* Hematologic malignancy
* QTc time prolongation >500 ms or history of familial long-QT-syndrome
* Heart failure NYHA III/IV
* Severe obstructive or restrictive ventilation disorder
* Concomitant use of known strong CYP3A Inhibitors
* Concomitant use of known strong CYP3A inducers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | At week 16 (after 5 cycles of study medication)
  Randomized, open-label, multicenter phase-II study comparing olaparib in combination with trabectedin versus physician's choice. Primary efficacy endpoint is the disease control rate after 5 cycles.

SECONDARY OUTCOMES:
Overall survival | Time from first administration of the IMP to time death from any cause until end of study (2.5 years)
  defined as the time from first administration of the IMP to time of death from any cause
Incidence of Treatment-Emergent Adverse Events | Time from first administration of the IMP to subjects end of trial (approximately month 6)
  This endpoint includes all AEs, their severity, SAEs, the relation of AEs to the study treatment, dose modifications for toxicity and discontinuation of study treatment during the trial phase. Toxic effects will be graded according to the National Cancer Institute Common Toxicity Criteria.
Patient reported outcomes | Before the first (week 0), at the third (week 8), and after the fifth treatment cycle (week 16)
  Patient reported outcomes (PROs) including health-related quality of life (QoL) are calculated as the new European Organization for Research and Treatment of Cancer (EORTC). QLQ-C30 summary score recommended by teh EORTC Quality of Life Group. In addition, the EORTC QLQ function and symptom scores are calculated according to the actual EORTC Scoring Manual.
Tumor response rate | At week 16 (after 5 cycles of study medication)
  Defined as the sum of complete remission (CR) and partial remission (PR) according to RECIST version 1.1 after 5 cycles of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Froehling, MD, Principal Investigator — NCT / DKFZ Heidelberg
Locations (9):
- Germany (9):
  - Medizinische Fakultät der TU Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - National Center for Tumordiseases (NCT), Heidelberg
  - Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München-Großhadern, München
  - Klinik Schillerhöhe, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided